CLINICAL TRIAL: NCT04309071
Title: Saliva Insulin Responses to a Standardized Meal Tolerance Test in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry); Core-Health Technologies Inc. (Unknown)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H18-02699
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Diet Modification; Insulin Resistance; Hyperinsulinemia
Keywords: Salivary insulin
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Salivary insulin responses to mixed meal tolerance test (Experimental): Saliva samples and finger prick glucose will be collected after at least 4 hours of fasting and then at 60 and 90 minutes following ingestion of a standardized meal tolerance test.
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — Salivary insulin responses to a standardized mixed meal

SUMMARY:
Recent evidence suggests that hyperinsulinemia (i.e., elevated insulin levels) is the primary causative factor in obesity. Insulin promotes fat storage and prevents fat breakdown, suggesting that weight loss would be optimized if insulin levels are managed and kept low. Understanding how different foods impact insulin levels could therefore aid in personalized weight loss (or weight maintenance) advice. It has been shown that salivary insulin can track plasma insulin following different meals and can delineate between lean and obese people. Thus, it was suggested that salivary insulin could be a potential surrogate for plasma insulin. The purpose of this study is to measure fasting saliva insulin, and salivary insulin responses to a standardized meal tolerance test in individuals with different body mass index (BMI).

ELIGIBILITY:
Inclusion Criteria:

* non-smoker
* have a body mass index greater than 18.5 kg/m2
* have not been diagnosed with type 2 diabetes or other medical conditions affecting glucose or insulin levels

Exclusion Criteria:

* You have been. diagnosed with diabetes (fasting blood sugar more than 7.0 mmol/l) or any other diagnosed chronic condition that may impact your glucose or insulin levels or the outcomes of this study.
* You take any medication which may affect your glucose and insulin level
* Unable to travel to make your testing appointments.
* Unable to consume the meal tolerance test drink/shake and/or provide finger stick glucose or saliva samples for the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Saliva insulin area under the curve | Measured for 90 minutes following the meal (time points: fasting, 60 minutes, and 90 minutes)
  The saliva insulin concentration measured by enzyme-linked immunosorbent assay - Area under the curve will be measured using the trapezoidal rule.
Saliva insulin at different time points | Salivary insulin at fasting (at least 4 hours of fasting), and at 60 and 90 minutes following mixed meal ingestion)
  Saliva insulin will be collected and measured by enzyme-linked immunosorbent assay.

SECONDARY OUTCOMES:
Glucose area under the curve | Measured for 90 minutes following the meal (time points: fasting, 60 minutes, and 90 minutes)
  Finger prick glucose concentration measured by glucometer - Area under the curve will be measured using the trapezoidal rule.
Glucose | Finger prick glucose will be measured at fasting (at least 4 hours of fasting), and at 60 and 90 minutes following mixed meal ingestion)
  Finger prick glucose at different time points will be measured by a glucometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No